CLINICAL TRIAL: NCT01129284
Title: The Treatment of Resistant Nephrotic Syndrome With ACTH Gel (ACTHAR)
Brief Title: Treatment of Resistant Nephrotic Syndrome With ACTH Gel (ACTHAR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Gerald B. Appel, Professor of Clinical Medicine, Nephrology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD9539
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-03

CONDITIONS: Treatment Resistant Nephrotic Syndrome
Keywords: Treatment Resistance; Nephrotic Syndrome; Focal Segmental Glomerulosclerosis; lipoid nephrosis; Membranous nephropathy; IgA nephropathy; proteinuria
MeSH Terms: conditions — Nephrotic Syndrome; Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Glomerulonephritis, Membranous; Glomerulonephritis, IGA; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acthar gel (Experimental): Patients will be treated with ACTHAR gel starting with 40 units given twice weekly subcutaneously for two weeks, then 80 units given twice weekly subcutaneously afterwards for a period of up to six months.
  Interventions: Drug: ACTHAR gel

INTERVENTIONS:
Drug: ACTHAR gel — Patients will be treated with ACTHAR gel starting with 40 units given twice weekly subcutaneously for two weeks, then 80 units given twice weekly subcutaneously afterwards for a period of up to six months.
  Other Names: H.P. Acthar gel

SUMMARY:
This study will examine the safety and effectiveness of ACTHAR Gel, when used to treat 15 patients diagnosed with "treatment resistant nephrotic syndrome."

Nephrotic syndrome is a group of symptoms that includes low levels of protein in the blood, swelling of tissue (edema), especially around the eyes, feet and hands; and high plasma levels of cholesterol. It is caused by a variety of diseases and underlying disorders that damage the kidneys, resulting in excessive excretion of protein in the urine. These diseases damage the glomeruli, which are small blood vessels that filter wastes and excess water from the blood and pass them into the bladder as urine. As a result of protein loss in the urine, the blood is deficient in protein. Normal amounts of blood protein are needed to help regulate fluid throughout the body. Protein in the blood normally draws water from the tissues and into the bloodstream. When blood protein levels are low, the normal movement of water is reversed, and fluid is drawn from the blood and accumulates in the tissues. This excess tissue fluid causes the swelling and puffiness (edema) that is a symptom of nephrotic syndrome.

Nephrotic syndrome is described as "treatment resistant" when a patient fails to achieve a sustained partial or complete remission after treatment with at least two first line therapies.

The goal of this study is to determine whether injections of ACTHAR Gel (an FDA approved treatment for nephrotic syndrome) over a six month period will lead to a correction of treatment resistant nephrotic syndrome in these patients.

DETAILED DESCRIPTION:
The nephrotic syndrome is characterized by heavy proteinuria, edema, hyperlipidemia, and a thrombotic tendency. Membranous nephropathy, focal segmental glomerulosclerosis, resistant minimal change disease, and Immunoglobulin A (IgA) nephropathy (also known as Berger's disease) are the common forms of idiopathic nephrotic syndrome in adults. Asymptomatic patients with idiopathic nephrotic syndrome may be treated with ACE inhibitors and /or angiotension receptor blockers to reduce proteinuria, with statins to treat hyperlipidemia, and diuretics to control edema.

Patients with large amounts of proteinuria are refractory to such treatments and often require immunosuppressive medications to promote a remission of the proteinuria and the nephrotic syndrome and to prevent progressive renal failure. All such immunosuppressives have multiple potential serious side effects. Some patients either relapse after remissions of their proteinuria or are resistant to immunosuppressive therapy.

A synthetic truncated analog of ACTH has been used in patients with the nephrotic syndrome in both uncontrolled trials and in a randomized controlled trial in membranous nephropathy. In uncontrolled studies it has led to sustained remissions of the nephrotic syndrome in multiple forms of idiopathic disease including membranous nephropathy and focal segmental glomerulosclerosis (FSGS). It has also led to reduction of total cholesterol, LDL cholesterol, Lpa, and elevations of HDL cholesterol. In a controlled randomized trial in membranous nephropathy it proved equivalent to an alternating monthly regimen of corticosteroids and an alkylating agent that is widely regarded as a first line therapy for this disease.

This synthetic truncated analog of ACTH is not available in the US. ACTHAR gel is a natural, highly purified, porcine ACTH which is both available in the US and FDA approved for use in the nephrotic syndrome. Although ACTHAR gel has been used to treat large numbers of patients with multiple sclerosis and infantile paralysis annually, it has, however, been used in only small numbers of patients for the indication of the nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Adult nephrotic patients, at least 18 years of age
2. Diagnosis of focal segmental glomerulosclerosis (FSGS), resistant or relapsing minimal change disease with failure to achieve a sustained partial or complete remission of the nephrotic syndrome after therapy with at least two first line therapies: corticosteroids and at least one other immunosuppressive regimen
3. Diagnosis of membranous nephropathy with failure to achieve a sustained partial or complete remission of the nephrotic syndrome after therapy with at least two first line therapies: either the "Ponticelli protocol" of alternating months of pulse steroids followed by oral steroids and then an alkylating agent with each regimen repeated for six full months of therapy or a calcineurin inhibitor, cyclosporine or tacrolimus, and at least one other therapy
4. Diagnosis of immunoglobulin A nephropathy (IgAN) with persistent nephrotic range proteinuria in patients on ACE inhibition or angiotension receptor blockers (ARB) therapy to reduce proteinuria
5. Willing and able to sign informed consent
6. Patients of childbearing age must agree to use birth control

Exclusion Criteria:

1. Patients under 18 years of age
2. Patients unable to sign informed consent
3. Patients having received rituximab or another monoclonal antibody within 6 months of the trial
4. Patients of childbearing age who refuse to use birth control
5. Patients with an estimated glomerular filtration rate (eGFR) less than 30 ml/min/1.73m2
6. Patients with other renal diseases (e.g. diabetic nephropathy, renal vascular disease) that would interfere with interpretation of the study.
7. Patients with comorbid conditions that would interfere with completion of the trial (malignancies, congestive heart failure (CHF), recent myocardial infarction).
8. Patients with known contraindications to the use of H.P. ACTHAR Gel, including: scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of a peptic ulcer, congestive heart failure, uncontrolled hypertension, and allergies to pork or pork products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald B Appel, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Bomback AS, Canetta PA, Beck LH Jr, Ayalon R, Radhakrishnan J, Appel GB. Treatment of resistant glomerular diseases with adrenocorticotropic hormone gel: a prospective trial. Am J Nephrol. 2012;36(1):58-67. doi: 10.1159/000339287. Epub 2012 Jun 19. PMID 22722778
- [Derived] Hogan J, Bomback AS, Mehta K, Canetta PA, Rao MK, Appel GB, Radhakrishnan J, Lafayette RA. Treatment of idiopathic FSGS with adrenocorticotropic hormone gel. Clin J Am Soc Nephrol. 2013 Dec;8(12):2072-81. doi: 10.2215/CJN.02840313. Epub 2013 Sep 5. PMID 24009220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 subjects with resistant glomerular diseases were enrolled and treated with ACTH gel (80 units subcutaneously twice weekly) for 6 months.
Groups:
- Membranous Nephropathy: Subjects diagnosed with membranous nephropathy were treated with ACTH gel (80 units subcutaneously twice a week) for 6 months.
- FSGS/MCD: Subjects diagnosed with focal segmental glomerulosclerosis (FSGS) or minimal change disease (MCD) were treated with ACTH gel (80 units subcutaneously twice a week) for 6 months.
- Immunoglobulin A (IgA) Nephropathy: Subjects diagnosed with Immunoglobulin A (IgA) nephropathy (Berger's disease) were treated with ACTH gel (80 units subcutaneously twice a week) for 6 months.
Period: Overall Study
Arm/Group | Membranous Nephropathy | FSGS/MCD | Immunoglobulin A (IgA) Nephropathy
Started | 5 | 5 | 5
Completed | 3 | 5 | 4
Not Completed | 2 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Membranous Nephropathy: Subjects diagnosed with membranous nephropathy
- FSGS/MCD: Subjects diagnosed with focal segmental glomerulosclerosis (FSGS) or minimal change disease (MCD)
- IgA Nephropathy: Subjects diagnosed with IgA nephropathy (Berger's disease)
- Total: Total of all reporting groups
Arm/Group | Membranous Nephropathy | FSGS/MCD | IgA Nephropathy | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 5 | 11
  >=65 years | 3 | 1 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 4 | 3 | 3 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 4 | 1 | 8
  African American | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 3 | 4
  Hispanic | 0 | 1 | 1 | 2
Previous Immunosuppressive therapy [Number; unit: participants]
  steroids | 0 | 0 | 2 | 2
  steroids, cyclosporine | 0 | 1 | 0 | 1
  steroids, cyclosporine, MMF | 0 | 1 | 0 | 1
  steroids, cyclosporine, tacrolimus | 1 | 1 | 0 | 2
  steroids, MMF | 0 | 0 | 1 | 1
  steroids, MMF, cyclophosphamide | 1 | 0 | 0 | 1
  steroids, tacrolimus | 0 | 1 | 0 | 1
  steroids, tacrolimus, cyclosporine, MMF | 0 | 1 | 0 | 1
  cyclosporine, MMF | 1 | 0 | 0 | 1
  MMF, cyclophosphamide | 1 | 0 | 0 | 1
  MMF, tacrolimus, cyclosporine, rituximab | 1 | 0 | 0 | 1
  none | 0 | 0 | 2 | 2
Renal Function [Number; unit: Participants]
  Impaired function: sCr range 1.6-2.9 mg/dl | 5 | 0 | 3 | 8
  Preserved function: sCr range 0.6-1.2 mg/dl | 0 | 5 | 0 | 5
  Preserved function: eGFR>60 ml/min/1.73m2 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Significant Reduction in Proteinuria to Remission Levels During the Treatment Period (Includes Complete and Partial Remission, as Defined in the Outcome Measure Description Below)
Description: Complete remission is defined as stable or improved renal function, serum creatinine < or = 125% baseline, with proteinuria falling <500 mg/day at month 6. Partial remission is defined as stable or improved renal function, serum creatinine < or = 125% baseline, with 50% reduction in proteinuria and final proteinuria 500-3500 mg/day at month 6.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Membranous Nephropathy: Subjects diagnosed with membranous nephropathy, treated with ACTH gel (80 units subcutaneously twice a week) for 6 months
- FSGS/MCD: Subjects diagnosed with focal segmental glomerulosclerosis (FSGS) or minimal change disease (MCD), treated with ACTH gel (80 units subcutaneously twice a week) for 6 months
- IgA Nephropathy: Subjects diagnosed with IgA nephropathy (Berger's disease), treated with ACTH gel (80 units subcutaneously twice a week) for 6 months
Arm/Group | Membranous Nephropathy | FSGS/MCD | IgA Nephropathy
Number analyzed (Participants) | 5 | 5 | 5
participants | 2 | 2 | 3

2. Secondary Outcome: Sustained Remissions up to 1 Year After Discontinuing Therapy
Description: Complete remission defined as stable or improved renal function, serum creatinine < or = 125% baseline, with proteinuria falling <500 mg/day at last follow-up visit (6 to 12 months post treatment). Partial remission defined as stable or improved renal function, serum creatinine < or = 125% baseline, with 50% reduction in proteinuria and final proteinuria 500-3500 mg/day at last follow-up visit (6 to 12 months post treatment).
Time Frame: Up to 1 year after treatment
Measure: Number; unit: participants
Arm/Group | Membranous Nephropathy | FSGS/MCD | IgA Nephropathy
Number analyzed (Participants) | 3 | 2 | 3
participants | 3 | 2 | 2

ADVERSE EVENTS:
Arm/Group | Membranous Nephropathy | FSGS/MCD | IgA Nephropathy
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Membranous Nephropathy (N=5) | FSGS/MCD (N=5) | IgA Nephropathy (N=5)
exacerbation of diabetes (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) — Subjects 1 and 2, both with membranous nephropathy (MN) and previous diagnoses of diet-controlled diabetes, had worsened glycemic control prompting initiation of oral hypoglycemic therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Membranous Nephropathy (N=5) | FSGS/MCD (N=5) | IgA Nephropathy (N=5)
Increased skin pigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — resolved within 4 weeks of discontinuing drug
Cushingoid response (General disorders) | 0 (0) | 0 (0) | 1 (1) — Cushingoid response: includes weight gain, Cushingoid facies, and increased blood pressure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes